CLINICAL TRIAL: NCT06046872
Title: Expanding Effective Report-back of Environmental Exposures Among New Researchers
Brief Title: Impacts of a Report-back Training Program
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Silent Spring Institute (Other)
Responsible Party: Principal Investigator, Jennifer Ohayon, Research Scientist, Silent Spring Institute
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 1R21ES032934-01A1 (NIH)
Record Dates: First submitted 2023-07-13; First posted 2023-09-21 (Actual); Last update posted 2025-05-18 (Actual); Status verified 2025-05

CONDITIONS: Behavioral Shift (Researcher Willingness to Report-back)

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Report-back training program (Other): Researchers participate in a training program on sharing personal results. Pre-and post-tests are administered to evaluate shifts in perspectives and wiliness to report-back before and after the training program. There is no control group.
  Interventions: Behavioral: Report-back training

INTERVENTIONS:
Behavioral: Report-back training — Researchers participate in a report-back training program to evaluate potential impacts on knowledge and future behaviors with respect to sharing personal exposure results with study participants.

SUMMARY:
Researchers participate in a hands-on training program on returning personal exposure results, and pre- and post-tests assess outcomes shifts in knowledge and perspectives on its value, and willingness to implement report-back in current or future studies.

DETAILED DESCRIPTION:
The investigators study the outcomes from a program that trains researchers to implement report-back, informs perspectives on the value of report-back, increases likelihood of adoption, and promotes insights from visualization of results. The investigators evaluate the training using pre- and post-tests. The training program includes an introductory module on ethical and practical benefits and best practices for report-back. This is followed by a session where researchers gain hands-on practice in report preparation using Digital Exposure Report-Back Interface (DERBI), a digital report-back tool. Pre- and post-tests assess outcomes related to their prior concerns about report-back, knowledge about report-back, shifts in perspectives on its value, novel insights about data from Researcher- DERBI, and willingness to implement report-back in current and future studies.

ELIGIBILITY:
Inclusion Criteria:

* Must be affiliated with a study that collects biomonitoring or personal exposure data

Exclusion Criteria:

* Under 18

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2023-06-22 (Actual); Primary Completion 2024-12-15 (Actual); Study Completion 2024-12-15 (Actual)

PRIMARY OUTCOMES:
Researcher wiliness to share personal exposure results as measured by pre- and post-tests administered alongside a training program | 3 hours (the training is approximately three hours and pre-and post-tests are administered directly before and after)
  Investigators are measuring if a training program on sharing personal exposure results impacts wiliness of other researchers to share personal results with participants in their current and future studies.

CONTACTS AND LOCATIONS:
Locations (1):
- Virtual and in-person across the U.S., Newton, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No